CLINICAL TRIAL: NCT06814262
Title: Effect of Clear Aligner Attachment Size on Extrusion of Maxillary Lateral Incisors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20031880
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Orthodontic Appliance Complication
Keywords: Extrusion of Maxillary Lateral Incisors; Clear Aligner Attachment

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control/optimized for extrusion.aligners (Placebo Comparator): The control will be Invisalign's optimized attachment which will be specifically optimized for extrusion.
  Interventions: Device: Corresponding treatment order in the prescription with Align Technology; Device: Superimposition of final and initial positions of lateral incisors: Predicted model
- Gingivally beveled 1x1x3mm aligners (Experimental): Each set of aligners would be worn for a week/gingivally beveled 1x1x3mm
  Interventions: Device: Corresponding treatment order in the prescription with Align Technology; Device: Superimposition of final and initial positions of lateral incisors: Gingivally beveled 1x1x3mm aligners
- Gingivally beveled 1x1x4mm aligners (Experimental): Each set of aligners would be worn for a week/gingivally beveled 1x1x4mm
  Interventions: Device: Corresponding treatment order in the prescription with Align Technology; Device: Superimposition of final and initial positions of lateral incisors: Gingivally beveled 1x1x4mm aligners
- Gingivally beveled 1x1x5mm aligners (Experimental): Each set of aligners would be worn for a week/gingivally beveled 1x1x5mm
  Interventions: Device: Corresponding treatment order in the prescription with Align Technology; Device: Superimposition of final and initial positions of lateral incisors: Gingivally beveled 1x1x5mm aligners

INTERVENTIONS:
Device: Corresponding treatment order in the prescription with Align Technology — Treating orthodontist placing the corresponding order in the prescription with Align Technology.
Device: Superimposition of final and initial positions of lateral incisors: Predicted model — Superimposition of final and initial positions of lateral incisors, two superimpositions will be completed. The pretreatment model will be superimposed with the predicted final model to establish the predicted movement of the maxillary lateral incisors
  Arms: Control/optimized for extrusion.aligners
Device: Superimposition of final and initial positions of lateral incisors: Gingivally beveled 1x1x3mm aligners — Superimposition of final and initial positions of lateral incisors, two superimpositions will be completed. The pretreatment model (Gingivally beveled 1x1x3mm aligners) will be superimposed with the posttreatment model to establish the actual movement of the maxillary lateral incisor.
  Arms: Gingivally beveled 1x1x3mm aligners
Device: Superimposition of final and initial positions of lateral incisors: Gingivally beveled 1x1x4mm aligners — Superimposition of final and initial positions of lateral incisors, two superimpositions will be completed. The pretreatment model (Gingivally beveled 1x1x4mm aligners) will be superimposed with the posttreatment model to establish the actual movement of the maxillary lateral incisor.
  Arms: Gingivally beveled 1x1x4mm aligners
Device: Superimposition of final and initial positions of lateral incisors: Gingivally beveled 1x1x5mm aligners — Superimposition of final and initial positions of lateral incisors, two superimpositions will be completed. The pretreatment model (Gingivally beveled 1x1x5mm aligners) will be superimposed with the posttreatment model to establish the actual movement of the maxillary lateral incisor.
  Arms: Gingivally beveled 1x1x5mm aligners

SUMMARY:
Orthodontic treatment has been revolutionized by clear aligner therapy, offering patients a more esthetic and comfortable alternative to traditional braces. In 1999, Align Technology introduced Invisalign. As Invisalign has increased in popularity and demand over the past two decades, clinical trials have shed light on the efficacy of Invisalign treatment. there have been changes in the Invisalign protocol such as introduction of SmartForce features in 2008, such as optimized attachments as well as the implementation of SmartTrack aligner material in 2011. Compared to conventional fixed orthodontic appliances, Invisalign cannot be adjusted on a visit-to visit basis. If ideal tooth movement has not been achieved after completion of the first sequence of aligners, additional trays, known as refinement trays, are required.

DETAILED DESCRIPTION:
There are various expert theories regarding the most effective methods of extrusion and multiple studies performed in vitro to evaluate the efficacy of different attachment types on the extrusion of lateral incisors, however only one in vivo clinical trial exists. There is a need for more randomized clinical trials that evaluate the effectiveness of different attachment designs for achieving optimal extrusion of lateral incisors. By determining the most effective attachment size for maxillary lateral incisor extrusion, this study can help improve treatment outcomes for orthodontic treatment with clear aligners and serve as a guide to assist clinicians in selecting the most effective attachment design.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with either Comprehensive Invisalign or Invisalign Teen treatment
* The maxillary arch has less than 6 mm of crowding or spacing
* Maxillary lateral incisors have a minimum of 0.3 mm of extrusion prescribed in the Tooth Movement Table on the Invisalign ClinCheck for the first set of aligners
* Maxillary lateral incisors within a normal range of bucco-lingual inclination
* Patients 12 years of age or older and either the patient or legal guardian are able to give consent
* Patients confirm good compliance throughout the study period

Exclusion Criteria:

* Patients do not complete all aligners in the first phase as prescribed
* Poor compliance recorded for aligner wear
* Restorations placed or oral surgery completed prior to final scan
* Midcourse intervention to improve tracking such as a bootstrap
* Maxillary lateral incisors not tracking and noted by minimum of 1 mm of aligner material incisally displaced when aligner fully seated
* Treatment plans include surgery or extractions
* Maxillary lateral incisors with pathology and restorations
* Missing teeth other than third molars
* Patients with anterior crossbite

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Determine which of three different attachment sizes offers more predictable extrusion of maxillary lateral incisors in subjects treated with clear aligners compared | baseline until the clear aligner treatment is completed at 20 to 25 weeks
  The aim of this prospective, randomized controlled trial is to determine which of three different attachment sizes (gingivally beveled 1x1x3 mm, gingivally beveled 1x1x4 mm, or gingivally beveled 1x1x5 mm) offers more predictable extrusion of maxillary lateral incisors in patients treated with clear aligners compared to control.

SECONDARY OUTCOMES:
Evaluate the accuracy of ClinCheck software | baseline until the clear aligner treatment is completed at 20 to 25 weeks
  To evaluate the accuracy of ClinCheck software in predicting the three-dimensional final position of the lateral incisor following extrusion using the attachment designs tested.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lindauer, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States